CLINICAL TRIAL: NCT04617743
Title: The Effect of Post-voiding Reisdual Urine on Non-muscle Invasive Bladder Cancer Recurrence and Progression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Mehmet Caglar Cakici, Department of Urology, Istanbul Medeniyet University
Other Study IDs: IMU Urology
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Bladder Cancer Recurrent; Non-Invasive Bladder Urothelial Carcinoma
Keywords: bladder cancer; post voiding residual urine; recurrence; non-muscle invasive bladder cancer; progression
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence; Non-Muscle Invasive Bladder Neoplasms; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High residual volume: Bladder tumor patients with high residual volume
- Low residual volume: Bladder tumor patients with low residual volume

SUMMARY:
Although transurethral resection is the main treatment option for stage Ta and T1 disease, relapse is frequently detected. Tumor number, tumor size, T stage, presence of in situ carcinoma and tumor grade are risk factors for recurrence. The relationship between post voiding residual urine volume and bladder tumor recurrence and progression has not been clearly established. The investigators aimed to examine the effect of high post voiding residual urine volume on recurrence and progression based on the hypothesis that tumor cells circulating in the bladder may increase with excess residual urine.

DETAILED DESCRIPTION:
Although transurethral resection is the main treatment option for stage Ta and T1 disease, relapse is frequently detected. Tumor number, tumor size, T stage, presence of in situ carcinoma and tumor grade are risk factors for recurrence. The relationship between post voiding residual urine volume and bladder tumor recurrence and progression has not been clearly established. Participants who underwent transurethral resection for bladder tumor will be included in the study. The investigators aimed to examine the effect of high post voiding residual urine volume on recurrence and progression based on the hypothesis that tumor cells circulating in the bladder may increase with excess residual urine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with transitional cell non-muscle invasive bladder cancer (NMIBC) pathology
* Patients with a diagnosis of Bladder cancer (NMIBC)
* Patients undergoing transurethral resection for bladder cancer (NMIBC)
* ≥18 years old patients

Exclusion Criteria:

* Non-transitional cell bladder cancers
* Patients with muscle-invasive bladder cancer pathology
* <18 years old patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with transitional cell non-muscle invasive bladder cancer pathology and patients with follow-up data
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 1 year
  Non-muscle invasive bladder cancer recurrence rate

SECONDARY OUTCOMES:
Progression | 1 year
  Non-muscle invasive bladder cancer progression rate

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Caglar Cakici, M.D., Principal Investigator — Istanbul Medeniyet University
Locations (3):
- Turkey (Türkiye) (3):
  - Health Sciences University, Dıskapi Yildirim Beyazit Training and Research Hospital, Ankara
  - Istanbul Medeniyet University, Istanbul
  - Health Sciences University, Tepecik Training and Research Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sazuka T, Sakamoto S, Nakamura K, Imamura Y, Yamamoto S, Komiya A, Ichikawa T. Impact of post-void residual urine volume on intravesical recurrence after nephroureterectomy for upper urinary tract urothelial carcinoma. Int J Urol. 2019 Dec;26(12):1106-1112. doi: 10.1111/iju.14103. Epub 2019 Sep 14. PMID 31522458
- [Result] Sazuka T, Sakamoto S, Imamura Y, Nakamura K, Yamamoto S, Arai T, Takeuchi N, Komiya A, Teishima J, Ichikawa T. Relationship between post-void residual urine volume, preoperative pyuria and intravesical recurrence after transurethral resection of bladder carcinoma. Int J Urol. 2020 Nov;27(11):1024-1030. doi: 10.1111/iju.14352. Epub 2020 Sep 1. PMID 32875619